CLINICAL TRIAL: NCT02313467
Title: Topical Application of 1.5% Butenyl ALA Without Light Source Irradiation in the Treatment of Acne: a Double Blinded Randomized Controlled Trial.
Brief Title: Topical PDT Cream Without Irradiation Source in the Acne Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNUH-PDT2
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Acne, Photodynamic Therapy
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.5% Butenyl ALA (Active Comparator): Topical application of 1.5% Butenyl ALA per every other day around acne lesions in the face
  Interventions: Drug: Topical application of 1.5% Butenyl ALA
- Control (Sham Comparator): Topical application of sham control per every other day around acne lesions in the face
  Interventions: Drug: Topical application of sham control

INTERVENTIONS:
Drug: Topical application of 1.5% Butenyl ALA
  Arms: 1.5% Butenyl ALA
Drug: Topical application of sham control
  Arms: Control

SUMMARY:
In this study, the investigators are going to compare the clinical effect and safety of topical application of 1.5% Butenyl ALA cream formula without light source irradiation in the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate acne vulgaris (Leeds revised acne grading system score 2-7) at baseline.

Exclusion Criteria:

* known pregnancy
* lactation
* any medical illness that might influence the results of the study
* a history of oral acne medication or surgical procedure, including laser treatment, within 6 months of study enrollment
* use of topical acne medication within 4 weeks of study enrollment.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percent change of inflammatory acne lesions compared with baseline | 12 week

SECONDARY OUTCOMES:
Percent change of non-inflammatory acne lesions compared with baseline | 12 week
Percent change of overall severity of acne lesions compared with baseline | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, MD, Principal Investigator — Seoul National University Department of Dermatology
Locations (1):
- Seoul National Unviersity, Seoul, Seoul Metropolitan, South Korea